CLINICAL TRIAL: NCT04324606
Title: A Phase I/II Study to Determine Efficacy, Safety and Immunogenicity of the Candidate Coronavirus Disease (COVID-19) Vaccine ChAdOx1 nCoV-19 in UK Healthy Adult Volunteers
Brief Title: A Study of a Candidate COVID-19 Vaccine (COV001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: COV001
Record Dates: First submitted 2020-03-20; First posted 2020-03-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Coronavirus
Keywords: COVID-19, Vaccine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — ChAdOx1 nCoV-19; MenACWY; Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (19):
- Group 1a (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19
  Interventions: Biological: ChAdOx1 nCoV-19
- Group 1b (Active Comparator): Volunteers will receive a standard single dose of MenACWY vaccine
  Interventions: Biological: MenACWY
- Group 1c (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 at week 0 and a boost dose of 5x10^10vp ChAdOx1 nCoV-19 9 months later
  Interventions: Biological: ChAdOx1 nCoV-19; Biological: ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) late vaccine (LV)
- Group 1d (Experimental): Volunteers will receive a standard single dose of MenACWY vaccine. 9 moths later they will receive two doses of 5x10^10vp ChAdOx1 nCoV-19 4-12 weeks apart
  Interventions: Biological: MenACWY; Biological: ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) late vaccine two (LVT)
- Group 2a (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19
  Interventions: Biological: ChAdOx1 nCoV-19
- Group 2b (Active Comparator): Volunteers will receive a standard single dose of MenACWY vaccine
  Interventions: Biological: MenACWY
- Group 2c (Experimental): Volunteers will receive two doses of 5x10^10vp ChAdOx1 nCoV-19 at week 0 and week 8
  Interventions: Biological: ChAdOx1 nCoV-19 full boost
- Group 2d (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 at week 0 and a boost dose of 2.5x10^10vp ChAdOx1 nCoV-19 at week 8
  Interventions: Biological: ChAdOx1 nCoV-19 half boost
- Group 2e (Active Comparator): Volunteers will receive two standard single doses of MenACWY vaccine at week 0 and week 8
  Interventions: Biological: MenACWY boost
- Group 2f (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 at week 0 and a boost dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x1010vp) a minimum of 4 weeks later
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL boost
- Group 2g (Active Comparator): Volunteers will receive two standard single doses of MenACWY vaccine a minimum of 4 weeks apart
  Interventions: Biological: MenACWY boost
- Group 3a (Experimental): Volunteers will receive one dose of 5x10^10vp ChAdOx1 nCoV-19 at week 0 and one dose of 5x10^10vp ChAdOx1 nCoV-19 at week 4
  Interventions: Biological: ChAdOx1 nCoV-19 full boost
- Group 3b (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 at week 0, a boost dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x1010vp) a minimum of 4 weeks later, and a third dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x1010vp) at 9 months
  Interventions: Biological: ChAdOx1 nCoV-19 full boost; Biological: ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) late vaccine (LV)
- Group 4a (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19
  Interventions: Biological: ChAdOx1 nCoV-19; Drug: Paracetamol
- Group 4b (Active Comparator): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 delivered intramuscularly
  Interventions: Biological: MenACWY; Drug: Paracetamol
- Group 4c (Experimental): Volunteers will receive a single dose of 5x10^10vp ChAdOx1 nCoV-19 at week 0 and a boost dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x1010vp) a minimum of 4 weeks later
  Interventions: Biological: ChAdOx1 nCoV-19; Biological: ChAdOx1 nCoV-19 0.5mL boost
- Group 4d (Active Comparator): Volunteers will receive two standard single doses of MenACWY vaccine a minimum of 4 weeks apart
  Interventions: Biological: MenACWY boost
- Group 5a (Experimental): Volunteers will receive two doses of 5x10^10vp ChAdOx1 nCoV-19 ≤ 16 weeks apart, and a third dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x1010vp) at 9 months
  Interventions: Biological: ChAdOx1 nCoV-19 full boost; Biological: ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) late vaccine (LV)
- Group 5b (Experimental): Volunteers will receive two standard single doses of MenACWY vaccine ≤ 16 weeks apart, a dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x1010vp) at 9 months then a second dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x1010vp) 4-12 weeks later
  Interventions: Biological: MenACWY boost; Biological: ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) late vaccine two (LVT)

INTERVENTIONS:
Biological: ChAdOx1 nCoV-19 — A single dose of 5x10^10vp of ChAdOx1 nCoV-19
  Arms: Group 1a; Group 1c; Group 2a; Group 4a; Group 4c
Biological: MenACWY — Standard single dose of MenACWY vaccine delivered intramuscularly
  Arms: Group 1b; Group 1d; Group 2b; Group 4b
Biological: ChAdOx1 nCoV-19 full boost — A single dose of 5x10^10vp of ChAdOx1 nCoV-19 followed by a boost dose of 5x10^10vp of ChAdOx1 nCoV-19
  Arms: Group 2c; Group 3a; Group 3b; Group 5a
Biological: ChAdOx1 nCoV-19 half boost — A single dose of 5x10^10vp of ChAdOx1 nCoV-19 followed by a boost dose of 2.5x10^10vp of ChAdOx1 nCoV-19
  Arms: Group 2d
Biological: MenACWY boost — A standard dose of MenACWY followed by a boost dose of MenACWY
  Arms: Group 2e; Group 2g; Group 4d; Group 5b
Drug: Paracetamol — 1g every 6 hours for 24 hours
  Arms: Group 4a; Group 4b
Biological: ChAdOx1 nCoV-19 0.5mL boost — A single dose of 5x10^10vp of ChAdOx1 nCoV-19 followed by a boost dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp)
  Arms: Group 2f; Group 4c
Biological: ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) late vaccine (LV) — A dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) 9 months after receiving a single or double dose of 5x10^10vp of ChAdOx1 nCoV-19
  Arms: Group 1c; Group 3b; Group 5a
Biological: ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) late vaccine two (LVT) — A dose of ChAdOx1 nCoV-19 0.5mL (3.5-6.5x10^10vp) 9 months after receiving a single or double dose of MenACWY, then a boost 4-12 weeks later
  Arms: Group 1d; Group 5b

SUMMARY:
A phase I/II single-blinded, randomised, multi-centre study to determine efficacy, safety and immunogenicity of the candidate Coronavirus Disease (COVID-19) vaccine ChAdOx1 nCoV-19 in UK healthy adult volunteers aged 18-55 years. The vaccine will be administered intramuscularly (IM) into the deltoid region of the arm

DETAILED DESCRIPTION:
There will be 4 study groups and it is anticipated that a total of 1090 volunteers will be enrolled. Volunteers will participate in the study for approximately 12 months from last vaccination visit (approximately 15 months from enrolment for participants receiving 2 doses)

ELIGIBILITY:
Inclusion Criteria

The volunteer must satisfy all the following criteria to be eligible for the study:

* Healthy adults aged 18-55 years.
* Able and willing (in the Investigator's opinion) to comply with all study requirements (participants must not rely on public transport or taxis).
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner and access all medical records when relevant to study procedures.
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination.
* Agreement to refrain from blood donation during the course of the study.
* Provide written informed consent.

Exclusion Criteria

The volunteer may not enter the study if any of the following apply:

* Planned receipt of any vaccine other than the study intervention within 30 days before and after each study vaccination .with the exception of the licensed seasonal influenza vaccination and the licensed pneumococcal vaccine. Participants will be encouraged to receive this vaccination at least 7 days before or after their study vaccine.
* Prior receipt of an investigational or licensed vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus vaccines).
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months, except topical steroids or short-term oral steroids (course lasting <14 days) .
* Any autoimmune conditions, except mild psoriasis, well-controlled autoimmune thyroid disease, vitiligo or stable coeliac disease not requiring immunosuppressive or immunomodulatory therapy.
* History of allergic disease or reactions likely to be exacerbated by any component of the ChAdOx1 nCoV-19 or MenACWY vaccines.
* Any history of angioedema .
* Any history of anaphylaxis .
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition likely to affect participation in the study (e.g. ongoing severe depression, history of admission to an in-patient psychiatric facility, recent suicidal ideation, history of suicide attempt, bipolar disorder, personality disorder, alcohol and drug dependency, severe eating disorder, psychosis, use of mood stabilisers or antipsychotic medication).
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
* Any other serious chronic illness requiring hospital specialist supervision.
* Chronic respiratory diseases, including mild asthma (resolved childhood asthma is allowed)
* Chronic cardiovascular disease (including hypertension), gastrointestinal disease, liver disease (except Gilberts Syndrome), renal disease, endocrine disorder (including diabetes) and neurological illness (excluding migraine)
* Seriously overweight (BMI≥40 Kg/m2) or underweight (BMI≤18 Kg/m2)
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Any clinically significant abnormal finding on screening biochemistry, haematology blood tests or urinalysis.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* History of laboratory confirmed COVID-19.
* New onset of fever or a cough or shortness of breath or anosmia/ageusia since February 2020. Should a reliable test become available, this exclusion criteria will be replaced with seropositivity for SARS-CoV-2 before enrolment.
* Those who have been at high risk of exposure before enrolment, including but not limited to: close contacts of confirmed COVID-19 cases, anyone who had to self-isolate as a result of a symptomatic household member, frontline healthcare professionals working in A&E, ICU and other higher risk areas. Should a reliable test become available, this exclusion criteria will be replaced with seropositivity for SARS-CoV-2 before enrolment.
* Living in the same household as any vulnerable groups at risk of severe COVID-19 disease (as per Public Health England guidance)

Additional exclusion criteria (subset of participants receiving Paracetamol in group 4 only)

• History of allergic disease or reactions likely to be exacerbated by Paracetamol

Re-vaccination exclusion criteria:

The following AEs associated with any vaccine, or identified on or before the day of vaccination constitute absolute contraindications to further administration of an IMP to the volunteer in question. If any of these events occur during the study, the subject will not be eligible to receive a booster dose and will be followed up by the clinical team or their GP until resolution or stabilisation of the event:

* Anaphylactic reaction following administration of vaccine
* Pregnancy. An exception to this will be prior to receipt of a booster dose at extra visit B. If a pregnant woman has discussed vaccination with their usual clinician (e.g. GP) and chooses to receive a COVID-19 vaccination, this may be administered by the trial team as part of extra visit B or as part of the provision of treatment to controls
* Any AE that in the opinion of the Investigator may affect the safety of the participant or the interpretation of the study results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1077 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Assess efficacy of the candidate ChAdOx1 nCoV-19 against COVID-19: Number of virologically confirmed (PCR positive) symptomatic cases | 6 months
  Number of virologically confirmed (PCR or NAAT positive) symptomatic cases of COVID-19
Assess the safety of the candidate vaccine ChAdOx1 nCoV: Occurrence of serious adverse events (SAEs) | Throughout the study, average of 18 months
  Occurrence of serious adverse events (SAEs) throughout the study until a cutoff date of 1st July 2021 or 6 months post late vaccination visit, whichever is latest

SECONDARY OUTCOMES:
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV: Occurrence of solicited local reactogenicity signs and symptoms | 7 days following vaccination
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following vaccination
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV: Occurrence of solicited systemic reactogenicity signs and symptoms | 7 days following vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following vaccination
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV: Occurrence of unsolicited adverse events (AEs) | 7 or 28 days following vaccination
  Occurrence of unsolicited adverse events (AEs) for 28 days following vaccination (7 days following vaccination for groups 1c, 1d, 5a & 5b)
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV through standard blood tests | 6 months
  Change from baseline for safety laboratory measures (haematology and biochemistry blood results)
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV by measuring the number of disease enhancement episodes | 6 months
  Occurrence of disease enhancement episodes
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 by hospital admissions | 6 months
  Number of hospital admissions associated with COVID-19
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 by ICU admissions | 6 months
  Number of intensive care unit admissions associated with COVID-19
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 by COVID-19 related deaths | 6 months
  Number of deaths associated with COVID-19
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 | 6 months
  Occurrence of severe COVID-19 disease (defined according to clinical severity scales)
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 by measuring seroconversion rates | 6 months
  Proportion of people who become seropositive for non-Spike SARS-CoV-2 antigens during the study
Assess cellular and humoral immunogenicity of ChAdOx1 nCoV-19 through ELISpot assays | 6 months
  Interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein
Assess cellular and humoral immunogenicity of ChAdOx1 nCoV-19 | 6 months
  Quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates)

OTHER OUTCOMES:
Assess cellular and humoral immunogenicity of ChAdOx1 nCoV-19 through Virus neutralising antibody assays | 6 months
  Virus neutralising antibody (NAb) assays against live and/or pseudotype SARS-CoV-2 virus
Assess safety, reactogenicity, immunogenicity and efficacy endpoints, for participants receiving prophylactic paracetamol | 6 months
  All safety, reactogenicity, immunogenicity and efficacy endpoints
Assess immunogenicity of ChAdOx1 nCoV-19 given as homologous prime-boost | 6 months
  Quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates) post boost
Compare viral shedding on stool samples of SARS-CoV-2 PCR or NAAT positive individuals | 6 months
  Differences in viral shedding on stool between vaccine and comparator arms at 7 days and beyond post SARS-CoV-2 PCR or NAAT positivity
Assess immunogenicity of a delayed three dose ChAdOx1 nCoV-19 schedule | Blood samples drawn at LV14, LV28 and LV182
  Quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates) post boost
assess immunological correlates of protection in relation to occurrence of COVID-19 disease in ChAdOx1 nCoV-19 recipients | Throughout the study, average of 18 months
  Immunological endpoints (antibody & cellular responses to SARS-COV2 spike protein) and COVID-19 disease endpoints (SARS-COV2 PCR positivity plus symptoms) in ChAdOx1 nCoV-19 recipients

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, Prof, Principal Investigator — University of Oxford
Locations (6):
- United Kingdom (6):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - St Georges University Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - CCVTM, University of Oxford, Churchill Hospital, Oxford
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Thomas TM, Hodgson SH, Emary K, Patrick-Smith M, Te Water Naude R, Stuart ASV, Henry J, English M, Moore M, Douglas N, Pollard AJ, Vanderslott S. The collective voice of early phase COVID-19 vaccine trial participants: Insights for improving confidence in novel vaccines. Hum Vaccin Immunother. 2023 Dec 31;19(1):2203023. doi: 10.1080/21645515.2023.2203023. PMID 37138460
- [Derived] Flaxman A, Marchevsky NG, Jenkin D, Aboagye J, Aley PK, Angus B, Belij-Rammerstorfer S, Bibi S, Bittaye M, Cappuccini F, Cicconi P, Clutterbuck EA, Davies S, Dejnirattisai W, Dold C, Ewer KJ, Folegatti PM, Fowler J, Hill AVS, Kerridge S, Minassian AM, Mongkolsapaya J, Mujadidi YF, Plested E, Ramasamy MN, Robinson H, Sanders H, Sheehan E, Smith H, Snape MD, Song R, Woods D, Screaton G, Gilbert SC, Voysey M, Pollard AJ, Lambe T; Oxford COVID Vaccine Trial group. Reactogenicity and immunogenicity after a late second dose or a third dose of ChAdOx1 nCoV-19 in the UK: a substudy of two randomised controlled trials (COV001 and COV002). Lancet. 2021 Sep 11;398(10304):981-990. doi: 10.1016/S0140-6736(21)01699-8. Epub 2021 Sep 1. PMID 34480858
- [Derived] Voysey M, Costa Clemens SA, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Clutterbuck EA, Collins AM, Cutland CL, Darton TC, Dheda K, Dold C, Duncan CJA, Emary KRW, Ewer KJ, Flaxman A, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Galiza E, Goodman AL, Green CM, Green CA, Greenland M, Hill C, Hill HC, Hirsch I, Izu A, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Libri V, Lillie PJ, Marchevsky NG, Marshall RP, Mendes AVA, Milan EP, Minassian AM, McGregor A, Mujadidi YF, Nana A, Padayachee SD, Phillips DJ, Pittella A, Plested E, Pollock KM, Ramasamy MN, Ritchie AJ, Robinson H, Schwarzbold AV, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, White T, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Single-dose administration and the influence of the timing of the booster dose on immunogenicity and efficacy of ChAdOx1 nCoV-19 (AZD1222) vaccine: a pooled analysis of four randomised trials. Lancet. 2021 Mar 6;397(10277):881-891. doi: 10.1016/S0140-6736(21)00432-3. Epub 2021 Feb 19. PMID 33617777
- [Derived] Barrett JR, Belij-Rammerstorfer S, Dold C, Ewer KJ, Folegatti PM, Gilbride C, Halkerston R, Hill J, Jenkin D, Stockdale L, Verheul MK, Aley PK, Angus B, Bellamy D, Berrie E, Bibi S, Bittaye M, Carroll MW, Cavell B, Clutterbuck EA, Edwards N, Flaxman A, Fuskova M, Gorringe A, Hallis B, Kerridge S, Lawrie AM, Linder A, Liu X, Madhavan M, Makinson R, Mellors J, Minassian A, Moore M, Mujadidi Y, Plested E, Poulton I, Ramasamy MN, Robinson H, Rollier CS, Song R, Snape MD, Tarrant R, Taylor S, Thomas KM, Voysey M, Watson MEE, Wright D, Douglas AD, Green CM, Hill AVS, Lambe T, Gilbert S, Pollard AJ; Oxford COVID Vaccine Trial Group. Phase 1/2 trial of SARS-CoV-2 vaccine ChAdOx1 nCoV-19 with a booster dose induces multifunctional antibody responses. Nat Med. 2021 Feb;27(2):279-288. doi: 10.1038/s41591-020-01179-4. Epub 2020 Dec 17. PMID 33335322
- [Derived] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Derived] Folegatti PM, Ewer KJ, Aley PK, Angus B, Becker S, Belij-Rammerstorfer S, Bellamy D, Bibi S, Bittaye M, Clutterbuck EA, Dold C, Faust SN, Finn A, Flaxman AL, Hallis B, Heath P, Jenkin D, Lazarus R, Makinson R, Minassian AM, Pollock KM, Ramasamy M, Robinson H, Snape M, Tarrant R, Voysey M, Green C, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 vaccine against SARS-CoV-2: a preliminary report of a phase 1/2, single-blind, randomised controlled trial. Lancet. 2020 Aug 15;396(10249):467-478. doi: 10.1016/S0140-6736(20)31604-4. Epub 2020 Jul 20. PMID 32702298